CLINICAL TRIAL: NCT06890923
Title: An Open Label, Multicenter Study of Nasal Foralumab in Non-Active Secondary Progressive Multiple Sclerosis Patients
Brief Title: Nasal Foralumab in Patients With Non-Active Secondary Progressive Multiple Sclerosis
Acronym: TILS-022
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tiziana Life Sciences LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IND 134155
Record Dates: First submitted 2025-02-12; First posted 2025-03-24 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-03

CONDITIONS: Non-Active Secondary Progressive Multiple Sclerosis
Keywords: Non-Active Secondary Progressive Multiple Sclerosis; Multiple Sclerosis; Foralumab; phase 2
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: All patients will initially receive nasal foralumab 50 µg three (3) days a week (Monday-Wednesday-Friday) for two weeks, followed by a one-week rest, comprising 3-week cycles. Patients meeting the requirements of the dose escalation rules will receive nasal foralumab 100 µg three (3) days a week (Monday-Wednesday-Friday) for two weeks, followed by a one-week rest, comprising 3-week cycles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nasal foralumab 50 μg per dosing day (25 μg per nostril) (Experimental): All patients will initially receive nasal foralumab 50 µg three (3) days a week (Monday-Wednesday-Friday) for two weeks, followed by a one-week rest, comprising 3-week cycles.
  Interventions: Drug: Foralumab TZLS-401 100 µg

INTERVENTIONS:
Drug: Foralumab TZLS-401 100 µg — Patients meeting the requirements of the dose escalation rules will receive nasal foralumab 100 µg three (3) days a week (Monday-Wednesday-Friday) for two weeks, followed by a one-week rest, comprising 3-week cycles.

SUMMARY:
Only subjects that have completed TILS-021, a Phase 2a Randomized, Double-Blind, Placebo-Controlled, Multicenter Dose-Ranging Study of Nasal Foralumab in Non-Active Secondary Progressive Multiple Sclerosis Patients are eligible to be enrolled in TILS-022. TILS-022 is a 6-month open-label extension study with an opportunity for dose to be escalated based on the subject's clinical status.

All subjects initiate dosing in this trial at a dose of nasal foralumab 50 µg 3 days a week (Monday, Wednesday, and Friday) for 2 weeks, followed by a 1-week rest, comprising a 3-week cycle. At week 12, the dose may be escalated to 100 µg according to pre-defined dose escalation rules. Study TILS-022 is intended to ensure all participants in TILS-021, a placebo-controlled study, will be able to receive open-label nasal foralumab for 6 months. The option to extend this trial for longer than 6 months will be explored with FDA by the Sponsor.

DETAILED DESCRIPTION:
TILS-021 (NCT06292923) is an ongoing Phase II dose-ranging study, the dosing regimen imitates that employed in the nonclinical studies that is, Monday-Wednesday-Friday for two consecutive weeks and then one rest week. This is believed to optimize the immunologic response to anti-CD3. It will assess the safety and potential efficacy as reflected in microglial activation on the PET scan, neurologic exam and measures, and immunologic changes in response to nasal foralumab administration in a randomized, double-blind, placebo-controlled, multicenter Phase II study of non-active secondary progressive MS patients with three months of treatment. Patients completing TILS-021will be eligible to enroll in study TILS-022. The primary objectives of this study in subjects with non-active secondary progressive multiple sclerosis (SPMS) that have successfully completed study TILS-022 are to evaluate 6-month (Day 169) safety data of nasal foralumab, as assessed by adverse event reports; changes in laboratory values; changes in physical, neurological, or nasal examinations; or changes in Total Nasal Symptom Score (TNSS). Objective 2 is to assess the clinical effect of foralumab after 6 months (Day 169) of treatment relative to baseline, as measured by the Modified Fatigue Impact Scale (MFIS).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have enrolled in and successfully completed TILS-021 within the preceding 90 days, including End of Treatment and End of Study assessments.
* Screening clinical laboratory studies are within the normal ranges or within the parameters specified below, and clinically acceptable in the opinion of the Investigator. Exceptions must be approved by the Clinical Research Organization or Sponsor's Medical Monitor.
* Adequate hematologic parameters without ongoing transfusion support:

  1. Hemoglobin (Hb) ≥ 9 g/dL
  2. Platelets ≥ 100 x 109 cells/L
* Creatinine ≤ 1.5 x the upper limit of normal (ULN), or calculated creatinine clearance ≥60 mL/minute x 1.73 m2 per the Cockcroft-Gault formula
* Total bilirubin ≤ 1.5 times the ULN unless due to Gilbert's disease.
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.0 times ULN.
* Negative urine pregnancy test within 7 days prior to the first dose of study therapy for women of childbearing potential, defined as a sexually mature woman who has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months (i.e., who has had menses any time in the preceding 24 consecutive months).
* Sexually active women of childbearing potential and male patients must agree to use two effective methods to avoid pregnancy (oral, injectable, or implantable hormonal contraceptives; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) throughout the study, and for 90 days after the completion of study treatment.
* Immunizations are current and up to date as adjusted for disease status and prior/current treatments and documented by the subject's treating neurologist.
* Ability and willingness to provide written informed consent.

Exclusion Criteria:

* Subjects that terminated TILS-021 early as defined as not undergoing an End of Treatment visit.
* Subjects that terminated TILS-021 early as defined as not undergoing an End of Study visit.
* Subjects that terminated TILS-021 due to any adverse events.
* Corticosteroid use (oral or intravenous) within the last 60 days or anticipated need for such treatment during the study period.
* Current use or use within 30 days prior to the Screening Visit of interferon, glatiramer acetate, fingolimod, siponimod, dimethyl fumarate, ponesimod, ozanimod, cyclosporin, methotrexate, azathioprine, mycophenolate mofetil, natalizumab or any other chronic immunosuppressive medication. Concomitant immunomodulatory or immunosuppressant treatments for MS are not permitted during study participation.
* Patient in whom the need to start or stop other pharmacologic treatment for MS is expected during the time of the study or the need for initiation of B cell depleting therapies (e.g.: ocrelizumab, ofatumumab, ublituximab, rituximab) during the study.
* Use of B cell depleting therapies (e.g.: ocrelizumab, ofatumumab, ublituximab, rituximab) at any time during study TILS-021 or after the patient has completed TILS-021 is not permitted.
* Subjects with any previous exposure to alemtuzumab, cyclophosphamide, cladribine, mitoxantrone, or daclizumab.
* Prior use of autologous hematopoietic stem cell transplantation or stem cell therapy.
* Nasal corticosteroids, nasal antihistamines, nasal flu dosing within the past 60 days.
* Active COVID-19 disease; according to FDA guidelines.
* Female patient who is pregnant, lactating, breastfeeding, or planning on becoming pregnant during the study. Female patients of childbearing age will undergo a serum pregnancy test at Screening, but prior to receiving their first dose, and be excluded from the study if positive. Urine pregnancy testing will be carried out prior to each dosing cycle, and the subject's study participation will be stopped if there is a positive result. Pregnancy testing will also be performed prior to each MRI imaging session and participation in the imaging session and the study will be terminated if positive.
* Any history of malignancy or active malignancy. This includes any skin cancers at any time.
* Inflammatory bowel disease, rheumatoid arthritis, systemic lupus erythematosus, asthma, or type 1 diabetes.
* Patients with a history of gadolinium allergy/contraindications or any other contraindications to MRI, such as metal implants, chronic renal disease and an eGRF of <30 mL/minute or claustrophobia. Or who are unable to lay flat in the PET or MRI scanner for the duration of the studies.
* Known positivity for human immunodeficiency virus, hepatitis B virus surface antigen (HBsAg), or hepatitis C virus or tuberculosis at Screening. If the subject has a history of positivity for any of these diseases, they are excluded even if current Screening is negative.
* Any nasal pathology such as clinically significant deviated septum, nasal polyps, chronic rhinitis, or a history of sinusitis diagnosed or treated in the past 12 months.
* Clinically significant cardiac condition or ECG abnormality at Screening or by history. An ECG will be done prior to each dosing cycle and patients will be excluded or treatment discontinued for any significant ECG abnormality.
* Any other medical intervention or other condition which, in the opinion of the Principal Investigator, could compromise adherence to study requirements or confound the interpretation of study results.
* Other than nasal foralumab, receipt of an investigational drug/biological product in the past 30 days of Screening, or concurrent receipt of an investigational drug during this study, other than the product under study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | Day 1 vs Day 169 (end of study)
  The safety and tolerability of 50 µg/dose and 100 µg/doses of foralumab nasal as measured by adverse event reports
Change in Baseline | Day 1 vs Day 169 (or termination)
  Assess change in baseline Modified Fatigue Impact Scale (MFIS) Scores range from 0-84. 0 is the minimum score and 84 is the maximum score. Lower scores indicate less fatigue while higher scores indicate increased fatigue.
Safety and Tolerability | Day 1 vs Day 169 (or termination)
  Blood pressure will be monitored at the beginning of every cycle. Increases and decreases in baseline will be monitored assessed for safety.
Safety and Tolerability | Day 1 vs Day 169 (or termination)]
  Heart rate will be monitored at the beginning of every cycle. Increases and decreases in baseline will be monitored assessed for safety.
Safety and Tolerability | Day 1 vs Day 169 (or termination)
  Lab values such as CHEM7 and CBC will be monitored at the beginning of every cycle on day 1. Any increases or decreases in baseline lab values will be assessed for safety.
Safety and Tolerability | Day 1 vs Day 169 (or termination)
  Total Nasal Symptom Score (TNSS). Scores range from 0-3 where 0 (minimum score) is no symptoms and 3 (maximum score) is severe. Higher scores indicate worse outcome.

SECONDARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue | Day 1 of study vs End of Study (Day 169) or Early Termination
  Assess change in baseline PROMIS Fatigue Short Form 7a. Scores range from 0-35 where the lower number indicated less fatigue.
Baseline Neurostatus Expanded Disability Status Scale (EDSS) | Day 1 of study vs End of Study (Day 169) or Early Termination.
  Assess change in baseline Neurostatus EDSS. Scores range from 0-10 where the lower number indicates less disability.
Baseline Multiple Sclerosis Functional Composite (MSFC-4) | Day 1 of study vs End of Study (Day 169) or Early Termination
  Assess change in baseline Multiple Sclerosis functional composite (MSFC-4)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided